CLINICAL TRIAL: NCT01914172
Title: Factors Affecting Health Promoting Behavior in Rare Disease Patients: A Mixed Methods Study of Men With Congenital Hypogonadotropic Hypogonadism (CHH)
Brief Title: Health Needs of Patients With Kallmann Syndrome
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Andrew Dwyer, Assistant Professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 233/13; 233/13 (Other: Commission Cantonale (Vaud))
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Kallmann Syndrome; Congenital Hypogonadotropic Hypogonadism; Idiopathic Hypogonadotropic Hypogonadism
Keywords: rare disease; community-based participatory research; health promotion; quantitative research; qualitative research; focus group
MeSH Terms: conditions — Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Online web-based questionnaire: Up to 200 patients with KS/CHH will be recruited to complete an online web-based questionnaire (less than 30 minutes to complete)
  Interventions: Other: online questionairres
- Patient focus group: Focus groups (90-120 minutes in duration) with 6-12 patients. Up to 36 patients total
- Online web-based evaluation of patient education materials: Up to 100 patients with KS/CHH will be recruited to complete an online web-based questionnaire to evaluate patient education materials (less than 15 minutes to complete)
  Interventions: Other: online questionairres

INTERVENTIONS:
Other: online questionairres — see group descriptions
  Other Names: patient focus groups
  Groups: Online web-based evaluation of patient education materials; Online web-based questionnaire

SUMMARY:
Kallmann syndrome (KS), also known as congenital hypogonadotropic hypogonadism (CHH), is a rare endocrine disorder that is characterized by failure to undergo puberty combined with infertility. KS/CHH patients face a number of psychosocial burdens related to delays in diagnosis, inadequate access to expert care, and lack of information about the condition. As such, there is some evidence to suggest that KS/CHH patients have unmet health needs. This study aims to identify the needs of patients and understand the issues that must be overcome to achieve improved health and quality of life.

DETAILED DESCRIPTION:
This study aims to examine the experiences of patients diagnosed with Kallmann syndrome (KS)/congenital hypogonadotropic hypogonadism (CHH).

The study includes two parts:

* online survey (less than 30 minutes to complete)
* focus groups with KS/CHH patients

The aim of this project is to better understand what health needs are not presently being met for these patients and to identify targets for improving the care of patients diagnosed with KS/CHH

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital hypogonadotropic hypogonadism: i.e. Kallmann syndrome or idiopathic hypogonadotropic hypogonadism
* Primary language is English/capable of responding to a written questionnaire in English
* Consenting to participate in the study

Exclusion Criteria:

* other diagnosis of hypogonadism: i.e. hypergonadotropic hypogonadism (Klinefelter syndrome), adult onset hypogonadism, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with congenital hypogonadotropic hypogonadism/Kallmann syndrome will be recuited internationally.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
illness perception | baseline
  subjective self-assessment questionnaire of how KS/CHH impacts a patient's life
depression symptoms | baseline
  self-rated questionnaire of depression symptoms
adherence to treatment | baseline
  self-report of adherence to medication treatment and periods without treatment or healthcare
understandability and actionability of patient education materials | baeline
  completion of Patient Education Materials Assessment Tool (PEMAT)

SECONDARY OUTCOMES:
coping | baseline
  Focus groups will be conducted to evaluate how KS/CHH impacts patients quality of life, the barriers to better health/quality of life, and how patients cope with living with KS/CHH
Interactions wth healthcare | baseline
  A questionnaire reporting the quality and type of interactions with healthcare providers and the healthcare system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dwyer, PhD, FNP-BC, Principal Investigator — Centre Hositalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Patient characteristics will be reported in aggregate (no identifiers)

REFERENCES:
- [Result] Dwyer AA, Quinton R, Morin D, Pitteloud N. Identifying the unmet health needs of patients with congenital hypogonadotropic hypogonadism using a web-based needs assessment: implications for online interventions and peer-to-peer support. Orphanet J Rare Dis. 2014 Jun 11;9:83. doi: 10.1186/1750-1172-9-83. PMID 24915927
- [Result] Dwyer AA, Quinton R, Pitteloud N, Morin D. Psychosexual development in men with congenital hypogonadotropic hypogonadism on long-term treatment: a mixed methods study. Sex Med. 2015 Mar;3(1):32-41. doi: 10.1002/sm2.50. PMID 25844173
- [Result] Dwyer AA, Tiemensma J, Quinton R, Pitteloud N, Morin D. Adherence to treatment in men with hypogonadotrophic hypogonadism. Clin Endocrinol (Oxf). 2017 Mar;86(3):377-383. doi: 10.1111/cen.13236. Epub 2017 Jan 11. PMID 27647266
- [Result] Dzemaili S, Tiemensma J, Quinton R, Pitteloud N, Morin D, Dwyer AA. Beyond hormone replacement: quality of life in women with congenital hypogonadotropic hypogonadism. Endocr Connect. 2017 Aug;6(6):404-412. doi: 10.1530/EC-17-0095. Epub 2017 Jul 11. PMID 28698240
- [Result] COST Action BM1105; Badiu C, Bonomi M, Borshchevsky I, Cools M, Craen M, Ghervan C, Hauschild M, Hershkovitz E, Hrabovszky E, Juul A, Kim SH, Kumanov P, Lecumberri B, Lemos MC, Neocleous V, Niedziela M, Djurdjevic SP, Persani L, Phan-Hug F, Pignatelli D, Pitteloud N, Popovic V, Quinton R, Skordis N, Smith N, Stefanija MA, Xu C, Young J, Dwyer AA. Developing and evaluating rare disease educational materials co-created by expert clinicians and patients: the paradigm of congenital hypogonadotropic hypogonadism. Orphanet J Rare Dis. 2017 Mar 20;12(1):57. doi: 10.1186/s13023-017-0608-2. PMID 28320476